CLINICAL TRIAL: NCT00146744
Title: Double-blind (Observer-blind), Randomised, Controlled, Phase I/II Study, to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Candidate Tuberculosis Vaccine, Mtb72F/AS02A Administered Intramuscularly at 0, 1, 2 Months to Healthy PPD-positive Volunteers Aged 18 to 50 Years
Brief Title: Safety and Immunogenicity of GSK Biological's Candidate Tuberculosis Vaccine Mtb72F/AS02A in Healthy PPD-positive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 102374
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis | interventions — Mtb72F-AS02A vaccine

INTERVENTIONS:
Biological: Mtb72F/AS02A

SUMMARY:
This study will evaluate the safety, reactogenicity and immunogenicity of Mtb72F/AS02A in healthy European volunteers who are PPD-positive either via previous vaccination with BCG and/or conversion to PPD positivity through exposure to Mycobacterium tuberculosis.

DETAILED DESCRIPTION:
The BCG vaccine has been widely available for several decades. It is easy and cheap to produce, and when given to neonates or young children it is effective in preventing severe manifestations of disease such as meningeal tuberculosis and miliary tuberculosis. However, in terms of the capacity of the vaccine to protect adult humans it shows a wide range of efficacy, including zero levels of protection. Due to the general realization that BCG is losing its protective effect, particularly in terms of preventing adult-onset tuberculosis, a major effort has been made to try to develop new alternative vaccines. One such candidate, Mtb72F/AS02A, is a polyprotein derived from two known M. tuberculosis antigens adjuvanted with AS02A. Mtb72F/AS02A is a candidate TB vaccine under development for two indications: prevention of primary TB infection in young children in highly endemic areas and as an adjunct to treatment for TB in adolescents and adults.

ELIGIBILITY:
INCLUSION CRITERIA

* Written informed consent
* Healthy PPD-positive volunteers aged 18 to 50 years
* No active pulmonary disease as confirmed by chest X-ray
* No history of extrapulmonary TB
* Seronegative for HIV 1 and 2, HBsAg, and HCV
* Clinically normal laboratory values for creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, complete blood count (CBC) and differential, haemoglobin, platelet count and urinalysis.
* Females : Non pregnant, must use adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

EXCLUSION CRITERIA

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* History of prior vaccination with experimental Mycobacterium Tuberculosis vaccines or experimental products containing MPL or QS21.
* Any confirmed or suspected immunosuppressive or immunodeficient condition; or family history of congenital or hereditary immunodeficiency.
* History of hypersensitivity to vaccines or vaccine components
* History of any acute or chronic illness or medication that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited symptoms during the 7-day follow-up period, unsolicited symptoms during the 30-day follow-up period, grade 3 vaccine related local and general symptoms during the 30-day follow-up and serious adverse events during the entire study

SECONDARY OUTCOMES:
Immunogenicity as assessed by humoral and CMI response.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lausanne, Switzerland

REFERENCES:
- [Derived] Spertini F, Audran R, Lurati F, Ofori-Anyinam O, Zysset F, Vandepapeliere P, Moris P, Demoitie MA, Mettens P, Vinals C, Vastiau I, Jongert E, Cohen J, Ballou WR. The candidate tuberculosis vaccine Mtb72F/AS02 in PPD positive adults: a randomized controlled phase I/II study. Tuberculosis (Edinb). 2013 Mar;93(2):179-88. doi: 10.1016/j.tube.2012.10.011. Epub 2012 Dec 5. PMID 23219236